CLINICAL TRIAL: NCT03899701
Title: Effective Use of PEC I, PEC II and Transversus Thoracics Muscle Plane Blocks for Subcutaneous Cardiac Pacemaker Insertion: A Case Series
Brief Title: Effective Use of Pecs and Transversus Thoracics Plane Blocks for Subcutaneous Cardiac Pacemaker Insertion: A Case Series
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never initiated and the PI has left the institution
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-9952
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEC I and PEC II block (Experimental): Ultrasound guided nerve block group.
  Interventions: Procedure: PEC I and PEC II blocks

INTERVENTIONS:
Procedure: PEC I and PEC II blocks — Participants will get a PEC I block with 10ml of 0.375% ropivacaine and a PEC II block with 20ml of 0.375% ropivacaine using ultrasound guidance.

SUMMARY:
Participants that undergo permanent cardiac pacemaker implantation can often present with challenging anesthetic management plans for the anesthesia provider. Typically, these procedures are performed in electrophysiology labs that are often in remote locations away from the main operating room suite. This presents the logistic challenges of not having standard anesthesia machines, equipment and medications readily available for these cases.Currently, the majority of these cases are done under local anesthesia with light to moderate sedation. However, when it comes to inserting more complex devices such as implantable cardiac defibrillators and cardiac resynchronization therapy devices, participants may not be able to tolerate these more invasive and painful procedures with only local anesthetic as the primary mode of analgesia.

Ultrasound-guided regional anesthetic techniques, in particular the pectoralis nerve blocks (PEC I and II) and the Transversus Thoracic Muscle plane block (TTP), offer an alternative mode of analgesia for these participants. PEC I blocks target the lateral and medial pectoral nerves by injecting local anesthetic in the fascial plane between the pectoralis major and minor muscles. PEC II blocks supplement the PEC I block by targeting the intercostal nerves with local anesthetic injected between the pectoralis minor and serratus anterior muscles. The transversus thoracic plane block targets the anterior cutaneous branches of the intercostal nerves. In combination, these four blocks would provide analgesia of the upper anterior chest wall.(3)These would provide effective analgesia of the upper anterior chest wall.(7).

However, there is a paucity of studies on the use of PEC blocks in cardiac pacemaker implantation procedures. There is a case report from 2014 on a 71 year-old male with an ejection fraction of 20% undergoing CRTD implantation, which showed that PECs block with moderate sedation using dexmedetomidine could be safely utilized to provide effective analgesia for the procedure.11 However, this was not a subcutaneous ICD that required tunneling of the coils. Thus there are no randomized controlled studies to investigate whether the use of peripheral nerve blocks as primary anesthetic choice could be a viable alternative for multiple participants undergoing subcutaneous ICD placement.

DETAILED DESCRIPTION:
This is a randomized controlled study evaluating the effectiveness of PEC I, PEC II, Transversus Thoracic plane blocks as the primary anesthetic in participants undergoing subcutaneous implantable defibrillator. There will be two groups; the nerve block group vs. general anesthesia group. The participants in the nerve block group will receive an ultrasound-guided nerve block in the electrophysiology suite prior to the start of the procedure. Participants will get a PEC I block with 10ml of 0.375% ropivacaine, PEC II block with 15ml of 0.375% ropivacaine, 15ml of 0.375% ropivacaine for TTP. PEC I block entails injecting local anesthesia between the pectoralis major and pectoralis minor muscles to anesthetize the medial and lateral pectoral nerves. PEC II block entails injecting local anesthetic between the pectoralis minor and serratus anterior muscles to block the upper intercostal nerves. For Tranversus Thoracic Plane block, local anesthetic will be injected between the internal intercostal muscle and the Transversus Thoracic muscle. The participants in the nerve block group will get mild sedation during the nerve blocks (midazolam 1-2mg IV and fentanyl 50-100mcg IV). After block placement, patient will be given a 0.3mcg/kg bolus of dexmedetomidine, then an infusion of dexmedetomidine 0.4mcg/kg/hr- 0.7mcg/kg/hr r +/- propofol 25mcg/kg/min-100mcg/kg/min for sedation. The general anesthesia group of participants will get the current standard of care with an endotracheal tube with a combination of IV induction medications and volatile anesthetic. Research assistant will hand an enclosed envelope to the anesthesiologists with the name of the group consented patient will be in.

Intraoperatively, the anesthesiologist will note if supplemental opioids and local anesthetic was required. Postoperatively, the PACU nurse will be asked to document pain scores according to the Visual Analog Scale (VAS) and total dose of opioids given. The distribution of the sensory block and motor weakness will be documented in the anesthesiologist's PACU discharge note. For postoperative data collection, opioid consumption totals and the pain scores at 30 minutes after arrival in PACU and at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing cardiac pacemaker placement Age 18 and above ASA II-IV

Exclusion Criteria:

* Patient refusal
* Inability to understand and sign consent
* Infection at the injection site
* Known allergy or hypersensitivity to ropivacaine or other amide local anesthetics
* Coagulopathy (INR > 1.5)
* Use of anticoagulant drugs that have not been discontinued in an appropriate amount of time before the surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Addition of local anesthetic by Interventionalist | within 4 hours
  The primary objective is to evaluate the utilization of perioperative rescue medications, including the supplementation of local anesthesia by the Internationalist.

SECONDARY OUTCOMES:
Presence of pain at the incision site at procedure start time | 20 minutes after block
  Presence of pain at the incision site at procedure start time
VAS Scores at 30 minutes after procedure and at discharge time | 30 minutes - 2 hours after procedure
  Comparison of VAS scores at 30 minutes after the procedure and at discharge time
Number of Patients with Prolong sensory deficit | 7 days after procedure
  Long-term follow-up (7 days) of prolong sensory deficit to the chest area
Use of Supplemental Opioid greater than 100mcg of Fentanyl | Within 4 hours
  The use of more than 100mcg of fentanyl by the anesthesiologists doing the case

CONTACTS AND LOCATIONS:
Overall Officials: Celina Joco, Study Director — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center- Wakefield Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable patient's data will be shared.

REFERENCES:
- [Background] Kaya E, Sudkamp H, Lortz J, Rassaf T, Janosi RA. Feasibility and safety of using local anaesthesia with conscious sedation during complex cardiac implantable electronic device procedures. Sci Rep. 2018 May 8;8(1):7103. doi: 10.1038/s41598-018-25457-x. PMID 29740019
- [Background] Kim DH, Kim S, Kim CS, Lee S, Lee IG, Kim HJ, Lee JH, Jeong SM, Choi KT. Efficacy of Pectoral Nerve Block Type II for Breast-Conserving Surgery and Sentinel Lymph Node Biopsy: A Prospective Randomized Controlled Study. Pain Res Manag. 2018 May 15;2018:4315931. doi: 10.1155/2018/4315931. eCollection 2018. PMID 29861803
- [Background] Fujiwara A, Komasawa N, Minami T. Pectoral nerves (PECS) and intercostal nerve block for cardiac resynchronization therapy device implantation. Springerplus. 2014 Aug 5;3:409. doi: 10.1186/2193-1801-3-409. eCollection 2014. PMID 25120950